CLINICAL TRIAL: NCT02397902
Title: Destiffening and Hypotensive Effects of Whole Milk and Full-fat Dairy Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Stephen J. Roy, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UTexasAustin
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Hypertension; Prehypertension
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dairy (Experimental): Add 4 daily servings of high fat dairy to diet for a period of 4 weeks
  Interventions: Dietary Supplement: High fat dairy
- Plant-based (Active Comparator): Add 4 daily servings of fruit to diet and/or plant-based milk, remove all dairy from diet for a period of 4 weeks
  Interventions: Dietary Supplement: Plant-based

INTERVENTIONS:
Dietary Supplement: High fat dairy — Add 4 daily servings per day of high fat dairy (yogurt, milk, cheese) for a period of 4 weeks
  Arms: Dairy
Dietary Supplement: Plant-based — Add 4 daily servings of fruit (fruit cup, apple sauce) and/or plant-based milk, remove all dairy for a period for 4 weeks
  Arms: Plant-based

SUMMARY:
The specific aim of the proposed study is to address the efficacy of conventional full-fat dairy products as part of the normal routine diet for improving vascular function and reducing blood pressure in middle-aged and older adults with elevated blood pressure. The investigators hypothesize that dietary intervention including whole milk and full-fat milk products will induce significant decreases in systolic blood pressure and arterial stiffness. The investigators also test the hypothesis that the reductions in blood pressure will be associated with the corresponding decreases in arterial stiffness and/or increases in endothelial vasodilatory function as well as improvements in arterial baroreflex sensitivity. If our hypotheses are supported by the results, the information could be used as a basis for recommendations for the use of whole milk and full-fat milk products in the secondary prevention of elevated blood pressure and vascular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Prehypertension or stage-1 hypertension

Exclusion Criteria:

* Consume > 3 servings of dairy or fruit per day
* Strenuous physical activity > 3 time per week
* Lactose intolerance, pregnancy, lactation, and/or alcohol abuse
* Taking cardiovascular-acting drugs
* Overt cardiovascular disease, metabolic disease, GI disorders and/or renal disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Seated blood pressure | 4 weeks

SECONDARY OUTCOMES:
24-hour ambulatory blood pressure | 4 weeks
Carotid arterial compliance as measured by arterial pressure and corresponding cross-sectional area by ultrasound | 4 weeks
Arterial stiffness as measured by pulse wave velocity between the aortic arch and femoral artery | 4 weeks
Flow mediated dilation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tanaka Hirofumi, PhD, Principal Investigator — The University of Texas at Austin; Stephen J Roy, MS, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States